

## Informed Consent/Authorization for Participation in Research

**Title of Research Study:** Phase I/II Study of PEGylated arginine deiminase (ADI-PEG20) with Carboplatin and Cabazitaxel in Men with Aggressive Variant Prostate Cancers (AVPC)

| <b>Study Number:</b> 2023-0467 | |
|--------------------------------|-----------------------|
| Principal Investigator: Ana Ap | aricio, MD |
| Participant's Name | Medical Record Number |

## **Key Information**

The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

# Why am I being invited to take part in a research study?

You are invited to take part in a research study because you have aggressive variant prostate cancer (AVPC).

# What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

# Why is this research being done?

The goal of this clinical research study is to find the best dose of ADI-PEG20 that can be given in combination with carboplatin and cabazitaxel to patients with AVPC.



This is an investigational study. ADI-PEG20 is not FDA approved or commercially available. It is currently being used for research purposes only. Carboplatin is FDA approved and commercially available for the treatment of ovarian cancer, but not for the treatment of AVPC. Cabazitaxel is FDA approved and commercially available for the treatment of prostate cancer that is metastatic (has spread). It is considered investigational to give ADI-PEG20 in combination with carboplatin and cabazitaxel to patients with AVPC.

The study doctor can explain how the study drugs are designed to work.

# How long will the research last and what will I need to do?

You may receive the study drugs for up to 2 years. Then every 6 months until the study ends or you withdraw from the study, the study staff will follow up with you to check on how you are doing.

You will be asked to visit the study clinic 1 time every week to receive the study drug(s) and have tests and procedures (such as physical exams, blood draws, imaging scans, and biopsies). Your samples (blood and tissue) will be used for routine tests and for research tests. The blood draws and biopsies collected for research purposes are not part of your standard care for the disease.

More detailed information about the study procedures can be found under "What happens if I agree to be in this research?"

# Is there any way being in this study could be bad for me?

Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. You should know that by taking part in this study, you may be forgoing standard-of-care treatment available for the disease. There may be FDA-approved treatments with established survival benefits for people with AVPC. You should discuss this with the study doctor.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

# Will being in this study help me in any way?

It cannot be promised that there will be any benefits to you or others from your taking part in this research. However, the study drugs may help to control the disease. Future patients may benefit from what is learned.



## What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

Instead of being in this research study, you may choose to receive chemotherapy (carboplatin and cabazitaxel) outside of this study. You may choose to receive other available standard of care treatment for the disease. You may receive other investigational therapy, if available. These alternative treatments have risks and benefits that may be the same or different than those in this research study. The study doctor can discuss these alternative treatments, including their risks and benefits, with you.

You may choose not to have treatment for cancer at all. If you decide that you don't want any more active treatment, one of your options is called "comfort care." Comfort care includes pain medication and other support. It aims to maintain your comfort and dignity rather than cure disease. Usually, this care can be provided at home. If you think you might prefer comfort care, please discuss this with your family, friends and your doctor.

In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

Your alternative to participating in this research study is to not participate.

# **Detailed Information**

The following is more detailed information about this study in addition to the information listed above.

# Who can I talk to if I have questions or concerns?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at 713-792-2830.

This research has been reviewed and approved by an Institutional Review Board (IRB – an ethics committee that reviews research studies). You may talk to them at 713-792-6477 or IRB Help@mdanderson.org if:

- Your questions, concerns, or complaints are not being answered by the research team
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.



## How many people will be in this study?

It is expected about 30 people at MD Anderson and MD Anderson Houston Area Locations will be enrolled in this research study.

## What happens if I agree to be in this research?

### Screening Tests

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an EKG to check your heart function.
- You will have a bone scan and then either an MRI, CT, or PET/CT scan to check the status of the disease.
- Blood (about 2½ tablespoons) will be drawn for:
  - Routine tests
  - Tumor marker testing. Tumor markers may be related to the status of the disease. The levels of tumor markers in your blood may indicate if the disease is getting worse or if the disease is responding to the study drugs. In this study, tumor markers include:
    - Prostate-specific antigen (PSA) level
    - Carcinoembryonic antigen (CEA) level
    - Prostatic acid phosphatase (PAP) level
    - Testosterone level
  - o Correlative research studies, which includes:
    - Anti-drug Antibody (ADA) testing ADA testing helps researchers learn if your immune system is making antibodies (proteins that attack foreign substances) against the study drug
    - Tests, including immune system tests and genetic tests, to better understand how the study drugs work and how they affect the tumor and levels of certain amino acids in the blood

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

#### **Study Groups**

If you are found to be eligible to take part in this study, you will be assigned to a study group and dose level of ADI-PEG20 based on when you join this study. Up to 2 dose levels of ADI-PEG20 may be tested. Up to 15 participants will be enrolled per dose level. The first group of participants will receive the lower dose level. The next group will receive the higher dose level, if no intolerable side effects are seen. One of these 2 doses will be selected as the best dose of ADI-PEG20 given in combination with carboplatin and cabazitaxel.



All participants will receive the same dose of carboplatin and cabazitaxel.

### **Study Drug Administration**

The study drugs are given in 2 phases: Induction Therapy and Maintenance Therapy. Each cycle of Induction Therapy is 21 days, and each cycle of Maintenance Therapy is 28 days.

### Induction Therapy (Cycles 1-6)

Induction Therapy is made of 6 study cycles:

- You will receive ADI-PEG20 as an injection into your muscle on Day -3 of Cycle 1 and then Days 1, 8, and 15 of Cycles 1-6. You will stay at the clinic for about 1 hour after each dose to be watched for side effects.
- You will receive cabazitaxel and carboplatin by vein over about 60 minutes each on Day 1 of Cycles 1-6.

On Day 1 when you receive all 3 study drugs, ADI-PEG20 will be given first. Then cabazitaxel will be given, followed by carboplatin.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

### Maintenance Therapy (Cycles 7 and beyond)

Starting at Cycle 7, you will receive only ADI-PEG20 as an injection into your muscle on Days 1, 8, 15, and 21 of Cycles 7 and beyond.

#### **Study Visits**

On Days -3, 8, and 15 of Cycle 1, and Days 1, 8, and 15 of each cycle thereafter, you will have some or all of the following tests:

- You will have a physical exam.
- Blood (up to 2½ tablespoons) will be drawn for routine tests, tumor marker testing, and/or correlative research studies.

**Before starting Cycles 1, 2, and 7**, you will have an image-guided tumor biopsy for correlative research studies. To perform an image-guided biopsy, a needle is inserted into the affected area using imaging such as CT, ultrasound, or MRI to collect cells or tissue from an organ, lymph node, or suspected tumor mass. The doctor will use the imaging to guide the needle into the area. Two (2) types of samples may be collected. It will either be a fine needle aspirate (FNA) that collects cells and/or a core biopsy that collects a small piece of tissue. This will be discussed with you.

**Every 3 cycles for up to 12 cycles and then every 4 cycles after that**, you will have a bone scan and then either an MRI, CT, or PET/CT scan to check the status of the disease. You may also have scan(s) at any time the study doctor thinks it is needed.



#### **End-of-Dosing Visit**

As soon as possible after your last dose of study drug(s):

- You will have a physical exam.
- Blood (about 2½ tablespoons) will be drawn for routine tests, tumor marker testing, and correlative research studies.
- You will have a bone scan and then either an MRI, CT, or PET/CT scan to check the status of the disease.

#### Follow-Up Visit

About 30 days after your last dose of study drug(s):

- You will have a physical exam.
- Blood (about 1 tablespoon) will be drawn for routine tests.

This visit may be done in person at the clinic or via a telemedicine appointment. Your blood sample may be collected at a local lab. The study staff will discuss this option with you.

#### Long-Term Follow-Up

Every 6 months after the Follow-Up Visit, the study staff will check on how you are doing. This information may be collected by calling you, scheduling a telemedicine appointment, or reviewing your medical records. If you are called or have a telemedicine appointment, it will take about 10 minutes. Long-term follow-up will continue until the study ends or you withdraw from the study.

#### Protocol PA13-0291

You will also be asked to take part in another research study: PA13-0291: Investigating Immunobiology in Cancer Patients. The goal of this study is to learn more about the immune cells (cells that the body makes to fight infection) of patients with cancer, and you will be asked to provide additional samples (such as blood, tissue, stool, urine, and/or oral/nasal samples). You will be given a separate consent form for this study, and it will be discussed with you in detail.

You must agree to participate in PA13-0291 in order to take part in this study. If you do not want to participate in PA13-0291, then you cannot take part in this study.

# What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for the following:

- Tell the study team about any symptoms or side effects you have, follow study directions, and come to all study appointments (or contacting the study team to reschedule).
- Tell the study doctor/study staff about all medications that you are taking or plan to take, including prescription and over-the-counter medications, supplements, vitamins, and herbal remedies.



You should not receive live virus and bacterial vaccines while you are receiving
the study drugs and for 30 days after your last dose of study drugs. Tell the study
doctor if you are planning to receive any vaccines during this time. They will
discuss with you if the type of vaccine is or is not allowed.

## What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you.

You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can then decide if you need to have any visits or tests to check on your health.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

# Is there any way being in this study could be bad for me? (Detailed Risks)

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

ADI-PEG20, carboplatin, and cabazitaxel each may cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia



and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

## **ADI-PEG20 Side Effects**

# Common (occurring in more than 20% of patients)

| fatigue | <ul> <li>injection site pain, redness, itching,</li> </ul> |
|---------|------------------------------------------------------------|
| | and/or skin rash |

## Occasional (occurring in 4-20% of patients)

| <ul> <li>headache</li> <li>dizziness</li> <li>mental status change</li> <li>difficulty sleeping</li> <li>fever</li> <li>chills</li> <li>hot flashes</li> <li>skin rash</li> </ul> | <ul> <li>mouth blisters/sores</li> <li>nausea/vomiting</li> <li>diarrhea</li> <li>constipation</li> <li>abdominal pain</li> <li>loss of appetite</li> <li>weight loss</li> <li>abnormal taste</li> <li>low blood cell counts</li> </ul> | <ul> <li>abnormal liver tests (possible liver damage)</li> <li>high blood levels of uric acid (possible painful joints and/or kidney failure)</li> <li>joint/muscle pain and/or swelling</li> <li>difficulty breathing</li> </ul> |
|---|---|---|
| <ul><li>skin rash</li><li>itching</li></ul> | <ul> <li>low blood cell counts<br/>(red, platelets, white)</li> </ul> | allergic reaction |

## Rare but serious (occurring in 3% of patients or fewer)

| • seizures | <ul> <li>immune system<br/>reaction (possible<br/>organ damage)</li> </ul> | life-threatening allergic<br>reaction (such as<br>difficulty breathing, low<br>blood pressure, and/or |
|---|---|---|
| | | organ failure) |

#### **Carboplatin Side Effects**

Common (occurring in more than 20% of patients)



| • | abnormal salts, |
|---|--------------------------|
| | minerals, and/or acids |
| | in the blood (possible |
| | weakness, swelling, |
| | fatigue, low blood |
| | pressure, organ |
| | failure, heart problems, |
| | changes in mental |
| | status, and/or seizure) |
| | • |

- vomiting
- low blood counts (red/white/platelets)
- pain

- abnormal liver tests (possible liver damage)
- abnormal kidney test (possible kidney damage)

### Occasional (occurring in 3-20% of patients)

| nerve damage |
|----------------------|
| (possible numbness, |
| pain, and/or loss of |
| motor function) |

- hair loss (partial or total)
- abdominal pain
- nausea
- constipation
- diarrhea

- weakness
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- infection

### Rare but serious (occurring in fewer than 3% of patients)

- high blood pressure
- dehydration
- destruction of red blood cells (possible anemia, kidney damage, and/or failure)
- blindness
- swelling of the eye nerve (possible vision loss)
- hearing loss
- kidney inflammation (possible kidney damage/failure)
- allergic reaction that may be lifethreatening (such as difficulty breathing, low blood pressure, and/or organ failure)

It is not known how often the following side effects may occur:

decreased bone marrow function

#### **Cabazitaxel Side Effects**

# Common (occurring in more than 20% of patients)

| fatigue | • vomiting | low blood cell counts |
|---|---|---|
| <ul><li>diarrhea</li></ul> | <ul><li>nausea</li></ul> | (red, platelets, white) |
| | <ul> <li>blood in the urine</li> </ul> | <ul><li>infection</li></ul> |

# Occasional (occurring in 3-20% of patients)



- swelling (arm/leg)
- irregular heartbeat
- low blood pressure (possible dizziness/fainting)
- fever
- dizziness
- headache
- hair loss (partial or total)
- loss of appetite
- abnormal taste

- dehydration
- constipation
- upset stomach
- abdominal pain
- weight loss
- mouth sores and/or blisters (possible difficulty swallowing)
- difficult and/or painful urination

- urinary tract infection
- nerve damage (possible numbness, pain, and/or loss of motor function)
- pain (back, joint, arm, leg, bone)
- muscle spasm
- weakness
- kidney failure
- difficulty breathing
- cough

### Rare but serious (occurring in fewer than 3% of patients)

- digestive system bleeding
- bladder inflammation (possible pain, bleeding, and/or urge to urinate)
- intestinal blockage
- hole in the intestines (possibly leaking contents into the abdomen)
- abnormal liver tests (possible liver damage and/or yellowing of the skin and/or eyes)
- lung inflammation (possible difficulty breathing)

## Frequency unknown

- changes in body salts such as sodium, potassium, and/or magnesium (possible fatigue and/or weakness)
- severe lifethreatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- severe allergic reaction (such as skin rash, skin redness, low blood pressure, and/or difficulty breathing due to a narrowing of the airways)

Receiving the study drug by vein may cause temporary irritation and/or bruising at the site of the infusion. It may also cause an allergic reaction.

# **Study Drug Combination Side Effects**

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.



#### **Other Risks**

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsy. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

A standard **bone scan** exposes you only to the radiation that comes from injecting the standard radioactive imaging solution for bone imaging.

During an **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

If an MRI contrast material is used, your study doctor will tell you about possible side effects or allergic reaction. Contrast agents can cause allergic reactions and kidney damage. Allergic reactions can include mild itching associated with hives but can also result in a serious life-threatening emergency from difficulty breathing. If this occurs, it is treatable. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an



uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

A PET scan may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort, or the scanning will be stopped. The PET scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

In addition to these risks, this research may hurt you in ways that are unknown. These may be a minor inconvenience or may be so severe as to cause death.

You will be told about any new information that may affect your health, welfare, or choice to stay in the research.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn baby, so you should not father a child while on this study.

**Birth Control Requirements:** If you can father a child and you are sexually active, you must use 1 form of highly effective birth control plus a barrier method (such as a condom) during the study and for 30 days after your last dose of ADI-PEG20. Talk to the study doctor about the birth control methods you should use during this study.

Tell the doctor right away if your partner becomes pregnant or suspects pregnancy during the study and for 30 days after your last dose of ADI-PEG20.

Do not donate sperm during the study and for 30 days after your last dose of ADI-PEG20.

# Will it cost anything to be in this study? Will I be paid to be in this study?

ADI-PEG20 will be provided at no cost to you during this study. You and/or your insurance provider will be responsible for the costs of carboplatin and cabazitaxel.



You and/or your insurance provider will not have to pay for certain research exams and procedures done that are covered by the study.

You and/or your insurance provider will be responsible for the costs of routine clinical services (such as diagnostic/therapeutic procedures, drugs, devices, laboratory assays, and other services that would ordinarily be ordered for medical care, regardless of whether or not you are participating in a study). There may be extra costs that are not covered by your medical plan that you will have to pay yourself.

Taking part in this study may result in added costs to you (such as transportation, parking, meals, or unpaid leave from work). You may have to pay for medication prescribed to treat or prevent side effects, and you may have to visit the clinic/hospital more often than if you were not participating in this study.

If you have insurance, talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this study. Also, find out if you need approval from your plan before you can take part in the study.

You may ask that a financial counselor be made available to you to talk about the costs of this study.

You will not receive any compensation for taking part in this study.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who need to review this information. Complete secrecy cannot be promised. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

A participant study number will be assigned to you once you have been enrolled in the study. This participant study number will be used to identify your data in the study report and when reporting any data from the study.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.



There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

The sponsor, monitors, auditors, the IRB, and the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access.

The results of this research may be published in scientific journals or presented at medical meetings. However, your identity will not be disclosed. Your name and other identifying information will be kept confidential.

Federal law provides additional protections of your medical records and related health information. These are described below.

# Will my data or samples be used for future research?

Your personal information and/or samples are being collected as part of this study. These data and/or samples may be used by researchers at MD Anderson, Polaris Group, and the National Institutes of Health, or shared with other researchers and/or institutions for use in future research.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the MD Anderson IRB before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research studies or shared with another researcher for future research studies without your additional informed consent.



## Can I be removed from the research study without my permission?

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

## What happens if I get hurt from being in this study?

If you get sick or hurt and it is related to your participation in this study, you will be given care at MD Anderson (if you are at the clinic when you are sick or hurt). If you get hurt or sick and you are not at the clinic (for example, you are at home or at another doctor's office):

- call your personal doctor right away (or in an emergency, call 911)
- tell your personal doctor or ER staff that you are in this study (try to give them a copy of this consent form or show them your participant card)
- call the study doctor (Dr. Ana Aparicio, at 713-792-2830) or 713-792-2121 (24 hours)

You will not be reimbursed for expenses or compensated financially by MD Anderson, Polaris Group, or the National Institutes of Health for this injury. Costs of treatment received because you were hurt or sick will be billed to you or your insurance company. No other form of payment is available.

You may also contact the MD Anderson IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

#### What else do I need to know?

This research is being sponsored and/or supported by Polaris Group and the National Institutes of Health.

MD Anderson may benefit from your participation and/or what is learned in this study.

Your information and samples (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will not contact you to let you know what they have found.



This research study involves genetic testing, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you.

The Genetic Information Nondiscrimination Act (GINA) prohibits health insurers or health plan administrators from requesting or requiring genetic information of you or your family members, or using such information for decisions regarding your eligibility for insurance or your premiums. However, this law does <u>not</u> provide the same protection for disability, life insurance, or long-term care insurance. GINA also prohibits most employers (with 15 employees or more) from using genetic information when making decisions on your employment, including decisions related to hiring, firing, promotion, pay, and job assignments. Please contact the study doctor if you would like more information about GINA and how it protects you from genetic discrimination.

Part of your care may be provided outside of MD Anderson by your home doctor(s).

## **Optional Procedures for the Study**

You do not have to agree to the optional procedures in order to take part in this study. There are no benefits to you for taking part in the optional procedures. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedures.

**Optional Procedure #1:** If you agree, you will have an image-guided tumor biopsy at the End-of-Dosing visit for correlative research studies. The study doctor will tell you what type of biopsy you will have and its risks.

**Optional Procedure #2:** If you agree, blood (about 2 tablespoons) will be drawn at the End-of-Dosing visit for correlative research studies. The study doctor will tell you what type of biopsy you will have and its risks.

### **Optional Procedure Risks**

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsy. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.



# CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have an image-guided tumor biopsy at the End-of-Dosing visit?

YES NO

**Optional Procedure #2:** Do you agree to have blood drawn for correlative studies at the End-of-Dosing visit?

YES NO

# Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Polaris Group and the National Institutes of Health, who is a sponsor or supporter of this study, and/or any future sponsors/supporters of the study, and/or licensees of the study technology
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will do its best to protect the privacy of your records, but it is possible that once information is shared with people listed on this form, it may be released to others. If this happens, your information may no longer be protected by federal law.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy



Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



## **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have about it, ask questions, and talk about it with others as need permission to enroll me on this study. By signing this conseany of my legal rights. I will be given a signed copy of this entropy of this entropy of the copy of this entropy. | ded. I give the study chair<br>ent form, I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| <u>WITNESS TO CONSENT</u> I was present during the explanation of the research to be μ protocol. | performed under this |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY A witness signature is only required for non-English speakers utilizing t short form consent process (VTPS) and patients who are illiterate. | |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSE | NT |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant an representative, using language that is understandable and have fully informed this participant of the nature of this stud and risks and that the participant understood this explanation | appropriate. I believe that I<br>ly and its possible benefits |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |



# **TRANSLATOR**

| nave translated the above informed consent as written (without additions or | | |
|---|---|---|
| subtractions) into | and assisted | and assisted the people |
| • | e of Language) | |
| obtaining and providing conscious consent process for this part | sent by translating all questions and resp<br>ticipant. | oonses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| | translator was a member of the researcl<br>an the translator, must sign the witness I | ` |